CLINICAL TRIAL: NCT04835155
Title: Faculty Member at Hasan Kalyoncu University
Brief Title: The Effect of The Premature Infant Oral Motorınterventıon on Suckıng Capacıty in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Selver Güler, Dr. Asst.Prof., Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Hasan Kalyoncu University
Record Dates: First submitted 2021-03-25; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Feeding Behavior; Premature Birth; Sucking Behavior
Keywords: Preterm Infant; Sucking Capacity; Premature Infant Oral Motor Intervention; Feeding; Oral Stimulation
MeSH Terms: conditions — Feeding Behavior; Premature Birth; Sucking Behavior

STUDY DESIGN:
Intervention Model Description: Sample The sample consisted of a total of 60 preterm infants all born after 26 weeks PMA with 30 each in the experimental and control group. Subjects were enrolled when they reached 29 or 30 weeks PMA and met inclusion criteria, and whose parents gave written consent.
  Random assignment to groups was performed by a research assistant, who was not involved in the research but worked in the same unit as the researchers, using the online software at https://www.randomizer.org. The primary nurses were blinded to groups, and the parents stepped out during therapy to assist in blinding.
Who Masked: Participant, Outcomes Assessor
Masking Description: The PIOMI was applied only by the trained researcher, and blind to the nursing staff in charge of care and feeding. No information about the PIOMI was shared with the general staff working in the NICU, and it was performed in the absence of the mothers, although no formal curtain was used for additional blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The researcher applied Premature Infant Oral Motor Intervention to the experimental group for 5 minutes per day for 14 consecutive days, 15-20 minutes before a sheduled feeding at either the 09:00 or 12:00 feeding. On the first day, the baseline sucking capacity of babies in experimental group was measured before any intervention. On the following 8th, 11th and 14th days, the measures of sucking capacity were repeated and followed by oral feeding trials. Growth measures were collected on the 1st and 14th days and the day of disharge.
  Interventions: Procedure: Premature Infant Oral Motor Intervention (PIOMI)
- control grup (No Intervention): The researcher did not apply any intervention. On the first day, the baseline sucking capacity of babies in control group was measured before any intervention. On the following 8th, 11th and 14th days, the measures of sucking capacity were repeated and followed by oral feeding trials.

INTERVENTIONS:
Procedure: Premature Infant Oral Motor Intervention (PIOMI) — The Premature Infant Oral Motor Intervention (PIOMI), developed by Dr. Brenda Lessen Knoll, was chosen for this study because it is the only oral motor program designed specifically for preterm babies as young as 29 weeks post menstrual age (PMA) and is the only program with a standardized training method and published intervention fidelity. The 5 minute therapy offers assisted movement to activate muscle contraction and movement against resistance to build strength in the perioral structures. The PIOMI has 8 steps where a provider uses a pinky finger to provide gentle stroking and pressure on the cheeks, lips, tongue, gums and palate to strengthen the oral sensory-motor functions and improve feeding efficiency. PIOMI ends with 2 minutes of NNS. NNS and oral stimulation have been found to mature the oral motor sensory system, and improve not only bottle feeding, but also breastfeeding.
  Arms: experimental group

SUMMARY:
ABSTRACT Objective: To test the effect of the Premature Infant Oral Motor Intervention (PIOMI) at 29-30 weeks post-menstrual age on the development of oral-motor function and sucking capacity.

Study Design: This study was a single-blind randomized controlled experimental design. The sample consisted of 60 preterm babies from two Neonatal Intensive Care Units in Gaziantep, Turkey between May 2019 and March 2020, with 30 each in the control and experimental groups. The PIOMI was applied to the experimental group for five minutes a day for 14 consecutive days. Sucking capacity, growth, feeding outcomes, and length of hospital stay (LOS) were measured. The Yakut Manometer Measuring Suction Power (PCT/TR2019/050678) was developed specifically for this study and tested for the first time.

DETAILED DESCRIPTION:
METHODS The data were obtained for 11 months between May 2019 and March 2020 in the NICUs of two different hospitals in the Gaziantep province of Turkey using a single-blind randomized controlled experimental design.

Eligibilty was determined by the neonatologist based on the following inclusion criteria: 1) babies born at 26-30 weeks PMA, 2) stable clinical condition, 3) vital signs stable for at least 24 hours, 4) able to have PIOMI by the 29th or 30th week PMA, 5) required respiratory support limited to an oxyhood, Continuous Positive Airway Pressure (CPAP) and/or nasal cannula up to 2L flow, 6) APGAR scores at 1- and 5-minutes of 4 and above, 7) any race or ethnicity, 8) intraventricular hemmorhage limited to level 1 or 2; and 9) had no birth defects including facial anomolies that would impact feeding.

Sample The sample consisted of a total of 60 preterm infants all born after 26 weeks PMA with 30 each in the experimental and control group. Subjects were enrolled when they reached 29 or 30 weeks PMA and met inclusion criteria, and whose parents gave written consent.

Random assignment to groups was performed by a research assistant, who was not involved in the research but worked in the same unit as the researchers, using the online software at https://www.randomizer.org. The primary nurses were blinded to groups, and the parents stepped out during therapy to assist in blinding.

Two subjects were lost during the research period. Subject number 15 in the experimental group died on the 11th day after enrollment of causes unrelated to the intervention. Subject number 31 in the control group was intubated on the 7th day after enrollment thus became ineligable. After a subject dropped out, the next subject enrolled replaced that subject and the study was continued with the same sample size.

Data Collection Tools The data were recorded on a Data Collection Form, a Follow-up Form for Daily Procedures Applied to the Infant, a Sucking Capacity Monitoring Form. The outcome measurements required preterm baby bottles and pacifiers, measuring tape for growth measurements, a scale, a bottle and pacifier sterilization machine, a labeling machine, and preterm baby silicone bottle nipples. Sucking capacity was measured by the Yakut Manometer Measuring Suction Power (Figure 1), a pressure manometer embedded into a silicone nipple developed specifically for this study by Prof. Dr. Yavuz Yakut (International Patent Number PCT/TR2019/050678). The PIOMI intervention required a stopwatch and infant monitors and no other equipment.

Ethical Approval Approval for this research was obtained and dated 9.03.2019 from Hasan Kalyoncu University Faculty of Health Sciences, Research Ethics Committee(2019/29). To ensure correct performance of the PIOMI, the researcher trained with Dr. Brenda Lessen Knoll, the founder of PIOMI, and competency was evaluated via review of a video-recording of the researcher doing PIOMI on a preterm baby (with written consent from the parents) using the Reliability Rating Tool (13) to ensure intervention fidelity. Written permission was received from Dr. Yakut to use his manometer for measuring sucking power in this study. Written informed consent was obtained from the parents of all subjects.

Test-Retest Reliability of the Manometer Measuring Suction Power To asses the reliability of the newly developed Yakut Manometer Measuring Suction Power it was tested on 10 preterm babies who had transitioned to full oral feedings and who had written consent from the parents and who were approved by a neonatologist. Each baby sucked on the manometer nipple for a minimum of one minute of successful sucking on two separate occcasions with a 5-minute interval in between. During both measurements, the highest value the infant could reach within the first minute after the baby began to suck was documented. The average sucking power at the 1st measure was 102±22.38 mmHg, and 104.5±13.83 mmHg at the 2nd measure. The test re-test reliability coefficient between the two applications was calculated by the Intraclass Correlation Coefficient (ICC) (2.1) and found to be 0.912. An ICC value of 0.75 indicates good reliability, and above .90 is excellent (33). The obtained ICC value of above 0.90 showed that the manometer was suitable / acceptable for use in clinical measurements (34).

Application Phase The PIOMI was applied only by the trained researcher, and blind to the nursing staff in charge of care and feeding. No information about the PIOMI was shared with the general staff working in the NICU, and it was performed in the absence of the mothers, although no formal curtain was used for additional blinding. Day 1 of the study was considered the 1st day that the babies received PIOMI. The researcher applied PIOMI to the experimental group for 5 minutes per day for 14 consecutive days, 15-20 minutes before a sheduled feeding at either the 09:00 or 12:00 feeding. On the first day, the baseline sucking capacity of babies in both groups was measured before any intervention. On the following 8th, 11th and 14th days, the measures of sucking capacity were repeated and followed by oral feeding trials. Growth measures were collected on the 1st and 14th days and the day of disharge (CONSORT Flow Diagram). A separate manometer nipple was used for each baby and labeled with names and surnames. Before each use, the bottle nipple was sterilized with a bottle and pacifier sterilization machine. Routine hand-washing was excercised before and after any patient or equipment contact. Babies were monitored during both the PIOMI application and the evaluation of the sucking capacity for any negative physiological/ behavioral cues of intolerance (apnea, bradycardia, desaturation below 90%, crying, tachycardia, facial color change). If one negative cue was observed, the procedure was suspended until the baby returned to normal, and was documented. The intervention would then be conitnued the following day.

ELIGIBILITY:
Inclusion Criteria:

Eligibilty was determined by the neonatologist based on the following inclusion criteria:

* babies born at 26-30 weeks PMA,
* stable clinical condition,
* vital signs stable for at least 24 hours,
* able to have PIOMI by the 29th or 30th week PMA,
* required respiratory support limited to an oxyhood, Continuous Positive Airway Pressure (CPAP) and/or nasal cannula up to 2L flow,
* APGAR scores at 1- and 5-minutes of 4 and above,
* any race or ethnicity,
* intraventricular hemmorhage limited to level 1 or 2; and
* had no birth defects including facial anomolies that would impact feeding.

Exclusion Criteria:

* Whose gestational age at birth was less than 26 weeks,
* had congenital disorder or birth trauma,
* had NEC,
* had RDS,
* were diagnosed with severe asphyxia,
* had intraventricular bleeding,
* had Newborn Withdrawal Syndrome,
* had Fetal Alcohol Syndrome,
* were receiving ventilator support,
* were receiving Extracorporeal Membrane Oxygenation,
* developed any complications during the follow-up period in the intervention group, whose balance status deteriorated,
* whose written and verbal permissions were obtained from their parents.

Ages: 29 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Baby's sucking power | The sucking power of the baby included in the study was measured up to 32 weeks.
  The suction power of the baby was measured in mmHg with the Manometer measuring the Sucking Power.
Baby's sucking before releasing the bottle | The sucking time without leaving the bottle of the baby included in the study was measured up to 32 weeks.
  The baby's sucking time without leaving the bottle was calculated in seconds.
Baby's total sucking time | The total sucking time of the baby included in the study was measured up to 32 weeks.
  The baby's total sucking time was calculated in seconds.
Baby's sucking amount | The sucking amount of the baby included in the study was measured up to 32 weeks.
  The baby's sucking amount was calculated in milliliters.

SECONDARY OUTCOMES:
Baby's body weight | The baby's body weight was measured for up to 40 weeks.
  Baby's body weight was measured in grams. height and head circumference.
Baby's height | Baby's height was measured for up to 40 weeks.
  Baby's height was measured in centimeters.
Baby's head circumference | Baby's head circumference was measured for up to 40 weeks.
  Head circumference of the baby was measured in centimeters.
First day of oral feeding time | The day when the baby was able to have the first oral feeding was measured up to 40 weeks.
  From the day the baby was included in the study, the day he sucked his mother was calculated. The average was calculated as 31 days in the experimental group and 41 days in the control group.
Discharge time | Up to 40 weeks were measured on the day of discharge.
  The total number of days the baby stayed in the hospital from the day he was included in the study was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Selver GÜLER, PhD, Principal Investigator — https://www.hku.edu.tr/
Locations (1):
- Hasan Kalyoncu University, Faculty of Health Sciences, Department of Nursing, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We plan to share it after it is ready for publication.

REFERENCES:
- [Result] Tian X, Yi LJ, Zhang L, Zhou JG, Ma L, Ou YX, Shuai T, Zeng Z, Song GM. Oral Motor Intervention Improved the Oral Feeding in Preterm Infants: Evidence Based on a Meta-Analysis With Trial Sequential Analysis. Medicine (Baltimore). 2015 Aug;94(31):e1310. doi: 10.1097/MD.0000000000001310. PMID 26252313
- [Result] Lessen Knoll BS, Daramas T, Drake V. Randomized Controlled Trial of a Prefeeding Oral Motor Therapy and Its Effect on Feeding Improvement in a Thai NICU. J Obstet Gynecol Neonatal Nurs. 2019 Mar;48(2):176-188. doi: 10.1016/j.jogn.2019.01.003. Epub 2019 Feb 2. PMID 30721652
- [Result] Fucile S, Gisel E, Lau C. Oral stimulation accelerates the transition from tube to oral feeding in preterm infants. J Pediatr. 2002 Aug;141(2):230-6. doi: 10.1067/mpd.2002.125731. PMID 12183719
- [Result] Lessen BS. Effect of the premature infant oral motor intervention on feeding progression and length of stay in preterm infants. Adv Neonatal Care. 2011 Apr;11(2):129-39. doi: 10.1097/ANC.0b013e3182115a2a. PMID 21730902
- [Result] Lessen BS, Morello CA, Williams LJ. Establishing Intervention Fidelity of an Oral Motor Intervention for Preterm Infants. Neonatal Netw. 2015;34(2):72-82. doi: 10.1891/0730-0832.34.2.72. PMID 26803089
- [Result] Kamitsuka MD, Nervik PA, Nielsen SL, Clark RH. Incidence of Nasogastric and Gastrostomy Tube at Discharge Is Reduced after Implementing an Oral Feeding Protocol in Premature (< 30 weeks) Infants. Am J Perinatol. 2017 May;34(6):606-613. doi: 10.1055/s-0037-1601443. Epub 2017 Apr 4. PMID 28376549
- [Result] Li XL, Liu Y, Liu M, Yang CY, Yang QZ. Early Premature Infant Oral Motor Intervention Improved Oral Feeding and Prognosis by Promoting Neurodevelopment. Am J Perinatol. 2020 May;37(6):626-632. doi: 10.1055/s-0039-1685448. Epub 2019 Apr 23. PMID 31013539
- [Result] Ghomi H, Yadegari F, Soleimani F, Knoll BL, Noroozi M, Mazouri A. The effects of premature infant oral motor intervention (PIOMI) on oral feeding of preterm infants: A randomized clinical trial. Int J Pediatr Otorhinolaryngol. 2019 May;120:202-209. doi: 10.1016/j.ijporl.2019.02.005. Epub 2019 Feb 5. PMID 30851536
- See also: Oral motor intervention improved the oral feeding in preterm infants: Evidence based on a meta-analysis with trial sequential analysis. — http://ncbi.nlm.nih.gov/pmc/articles/PMC4616601/
- See also: Effect of the premature infant oral motor intervention on feeding progression and length of stay in preterm infants. — https://journals.lww.com/advancesinneonatalcare/Abstract/2011/04000/Effect_of_the_Premature_Infant_Oral_Motor.12.aspx
- See also: Establishing intervention fidelity of an oral motor intervention for preterm infants. — https://www.researchgate.net/publication/282553446_Establishing_Intervention_Fidelity_of_an_Oral_Motor_Intervention_for_Preterm_Infants
- See also: Incidence of nasogastric and gastrostomy tube at discharge is reduced after implementing an oral feeding protocol in preterm (<30 weeks) infants. — https://www.thieme-connect.com/products/ejournals/abstract/10.1055/s-0037-1601443
- See also: Early premature infant Oral motor intervention improved oral feeding and prognosis by promoting neurodevelopment. — https://www.thieme-connect.com/products/ejournals/abstract/10.1055/s-0039-1685448